CLINICAL TRIAL: NCT00550680
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety, and Tolerability of Once-Monthly Administration of Intravenous C.E.R.A. for the Maintenance of Haemoglobin Levels in Dialysis Patients With Chronic Renal Anaemia
Brief Title: A Study of Mircera for the Maintenance Treatment of Participants With Chronic Renal Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20952; 2006-006349-15 (EudraCT Number)
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Renal Anemia
MeSH Terms: interventions — continuous erythropoietin receptor activator

ARMS (1):
- Mircera in Renal Anemia (Experimental): Participants with chronic renal anemia who have been previously treated with erythropoiesis-stimulating agent (ESA) therapy will receive IV Mircera every 4 weeks for a total of 24 weeks in this single-arm study. The first dose of 120, 200, or 360 mcg will be determined by the dose of ESA received prior to administration of study treatment. Subsequent doses will be adjusted to maintain Hb concentrations within target of 10.5 and 12.5 grams per deciliter (g/dL).
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta — Participants will receive a starting dose of 120, 200, or 360 mcg via IV injection. Thereafter, the once-monthly dose will be titrated to achieve target Hb concentrations.
  Other Names: Mircera/CERA

SUMMARY:
This single-arm study will assess the efficacy and safety of intravenous (IV) Mircera when administered for the maintenance of hemoglobin (Hb) levels in participants with chronic renal anemia. Individuals currently receiving maintenance treatment with epoetin alfa or darbepoetin alfa will receive monthly injections of Mircera, with the starting dose (120, 200, or 360 micrograms [mcg] IV injection) derived from the dose of epoetin alfa or darbepoetin alfa they were receiving in the week preceding study start.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age
* Chronic renal anemia
* Stable epoetin alfa or darbepoetin alfa therapy for past 2 months
* Hemodialysis therapy for ≥3 months

Exclusion Criteria:

* Transfusion of red blood cells during previous 2 months
* Poorly controlled hypertension requiring hospitalization or interruption of ESA treatment in previous 6 months
* Acute or chronic bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Greece (14):
  - Aigáleo
  - Athens
  - Corinthos
  - Daphni-athens
  - Ioannina
  - Kalamata
  - Kyparissía
  - Lamia
  - Larissa
  - Livadeia
  - Mytilene
  - Pátrai
  - Rhodes
  - Thessaloniki

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera in Renal Anemia: Participants with chronic renal anemia who were previously treated with erythropoiesis-stimulating agent (ESA) therapy received intravenous methoxy polyethylene glycol-epoetin beta (Mircera), also known as continuous erythropoietin receptor activator (CERA), every 4 weeks for a total of 24 weeks in this single-arm study. The first dose of 120, 200, or 360 micrograms (mcg) was based upon the dose of ESA received prior to administration of study treatment, while subsequent doses were adjusted to maintain hemoglobin (Hb) concentrations within target of 10.5 and 12.5 grams per deciliter (g/dL).
Period: Overall Study
Arm/Group | Mircera in Renal Anemia
Started | 208
Completed | 152
Not Completed | 56
Not completed — Administrative Reasons | 1
Not completed — Adverse Event | 5
Not completed — Death | 3
Not completed — Early Improvement | 1
Not completed — Lost to Follow-up | 3
Not completed — Lack of Efficacy | 1
Not completed — Other | 10
Not completed — Protocol Violation | 7
Not completed — Refused Treatment | 19
Not completed — Screen Failure | 6

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of Mircera/CERA and had at least one safety follow-up assessment.
Groups:
- Mircera in Renal Anemia: Participants with chronic renal anemia who were previously treated with ESA therapy received intravenous Mircera/CERA, every 4 weeks for a total of 24 weeks in this single-arm study. The first dose of 120, 200, or 360 mcg was based upon the dose of ESA received prior to administration of study treatment, while subsequent doses were adjusted to maintain Hb concentrations within target of 10.5 and 12.5 g/dL.
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (14.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 115

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Average Hb Within Plus/Minus (±) 1 g/dL of Reference Hb and Within Target Range During the Efficacy Evaluation Period (EEP)
Description: Reference Hb was determined individually per participant as the average of all Hb values during a pre-treatment stability assessment (Weeks -4 to 0). During the EEP (Weeks 17 to 24), participants provided a total of four blood samples for Hb monitoring while on treatment with Mircera/CERA. The average Hb during the EEP was calculated per participant and assessed against the reference value. The percentage of participants who had average Hb during the EEP in the target range of 10.5 to 12.5 g/dL and within ±1 g/dL of their individual reference Hb was determined as the primary endpoint. The 95 percent (%) confidence interval (CI) was calculated using the Pearson-Clopper method for exact confidence bounds.
Time Frame: Weeks -4, -3, -2, -1,and 0; pre-dose (0 hours) during Weeks 18, 20, 22, and 24
Population: Per Protocol (PP) Population: All participants who received at least one dose of Mircera/CERA and provided data for at least one follow-up assessment, and who fulfilled inclusion/exclusion criteria per study protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 149
percentage of participants | 53.7 [45.4 to 61.9]

2. Secondary Outcome: Mean Change in Time-Adjusted Hb From Baseline to EEP
Description: Reference Hb was determined individually per participant as the average of all Hb values during a pre-treatment stability assessment (Weeks -4 to 0). During the EEP (Weeks 17 to 24), participants provided a total of four blood samples for Hb monitoring while on treatment with Mircera/CERA. The average Hb during the EEP was calculated per participant and assessed against the reference value. The mean change in Hb value between reference (i.e., "Baseline") Hb and the EEP average Hb was calculated and expressed in g/dL.
Time Frame: At Weeks -4, -3, -2, -1, and 0; pre-dose (0 hours) during Weeks 18, 20, 22, and 24
Population: Intent-to-Treat (ITT) Population: All participants who received at least one dose of Mircera/CERA and provided data for at least one follow-up assessment.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 187
g/dL | 0.0 (1.17)

3. Secondary Outcome: Percentage of Participants Whose Hb Remained Within Target Range Throughout the EEP
Description: During the EEP (Weeks 17 to 24), participants provided a total of four blood samples for Hb monitoring while on treatment with CERA/Mircera. The percentage of participants who maintained each single Hb measurement in the target range of 10.5 to 12.5 g/dL was determined. The 95% CI was calculated using the Pearson-Clopper method for exact confidence bounds.
Time Frame: Pre-dose (0 hours) during Weeks 18, 20, 22, and 24
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 187
percentage of participants | 53.7 [46.3 to 61.0]

4. Secondary Outcome: Mean Time Spent in the Target Range for Hb During the EEP
Description: During the EEP (Weeks 17 to 24), participants provided a total of four blood samples for Hb monitoring while on treatment with Mircera/CERA. Time spent in the target range of 10.5 to 12.5 g/dL was defined as time from first on-target Hb to time of last known on-target Hb, as collected during the EEP. Time spent in the target range was averaged among all participants and expressed in days.
Time Frame: Pre-dose (0 hours) during Weeks 18, 20, 22, and 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 187
days | 34 (18.1)

5. Secondary Outcome: Percentage of Participants Who Required Any Dose Adjustment of Mircera/CERA During the Dose Titration Period (DTP) and EEP
Description: Study drug administration occurred monthly during the DTP (Weeks 0 to 16), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during Week -1. Subsequent doses could be adjusted throughout the study including during the EEP (Weeks 17 to 24) on the basis of Hb levels or other modification criteria. The percentage of participants who required a dose adjustment for any reason was calculated during the DTP and EEP.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; number (n) of participants who entered each treatment period was reported.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 187
percentage of participants
  DTP (n=187) | 68
  EEP (n=160) | 38

6. Secondary Outcome: Number of Participants Prematurely Withdrawn From the Study to Receive Blood Transfusion
Description: The number of participants who were prematurely withdrawn from the study to receive a blood transfusion during treatment, including the DTP (Weeks 0 and 16) and/or EEP (Weeks 17 to 24), was reported.
Time Frame: Continuously and at every visit from Week 0 (every week until Week 2, thereafter every 2 weeks) through Week 24
Population: All Enrolled Population: Includes all participants enrolled into the study regardless of treatment received.
Measure: Number; unit: participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 208
participants | 3

ADVERSE EVENTS:
Time Frame: Continuously and at every visit from Week -4 (every week until Week 2, every 2 weeks until Week 24) through Week 28
Description: Safety Population
Arm/Group | Mircera in Renal Anemia
Serious Adverse Events (participants affected / at risk) | 34/188
Other Adverse Events (participants affected / at risk) | 10/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera in Renal Anemia (N=188)
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac valve disease (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Arteriovenous graft site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Obstructive uropathy (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Amputation (Surgical and medical procedures) | 1
Nephrectomy (Surgical and medical procedures) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera in Renal Anemia (N=188)
Hypertension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.